CLINICAL TRIAL: NCT00871325
Title: Effect of Gastrointestinal Nerve Modulation With DAIKENCHUTO (TU-100) on Gastrointestinal and Colonic Transit in Humans
Brief Title: Effect of TU-100 on Gastrointestinal and Colonic Transit in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: TU100CPT1
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Postoperative Ileus
Keywords: Gastric emptying; Small bowel transit; Colonic transit; Whole gut transit; Postoperative Ileus
MeSH Terms: interventions — dai-kenchu-to; 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daikenchuto (TU-100) 7.5g/day (Experimental): Daikenchuto (TU-100) 2.5g TID (7.5g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Daikenchuto (TU-100) 15g/day (Experimental): Daikenchuto (TU-100) 5g TID (15g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Placebo (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daikenchuto (TU-100) — Subjects will receive 2.5g TID (7.5g/day) of TU-100. Dosage form is a granule. Subject will take a daily dose divided three times a day for 5 days.
  Arms: Daikenchuto (TU-100) 7.5g/day
Drug: Daikenchuto (TU-100) — Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is a granule. Subject will take a daily dose divided three times a day for 5 days.
  Arms: Daikenchuto (TU-100) 15g/day
Drug: Placebo — Subjects will receive daily dose of TU-100 placebo. Dosage form is a granule. Subject will take a daily dose divided three times a day for 5 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the dose related effects of orally administered TU-100, a botanical agent that modulates gastrointestinal nerves, on gastrointestinal motility and colonic transit of solids.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent
* Males and non-pregnant, non-breastfeeding females;
* Subject is willing to undergo multiple radionuclide scans
* Subject BMI is between 18 and 35 kg/m2
* Subject has a negative urine drug screen
* Subject has screening laboratory values that are within normal range for the analyzing laboratory

Exclusion Criteria:

* Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders.
* Unable to withdraw medications 48 hours prior to the study:
* Alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, SSRI and newer antidepressants.
* Analgesic drugs including opiates, NSAID, COX 2 inhibitors
* GABAergic agents
* Benzodiazepines

NOTE: Low stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection and birth control pills or depot injections are permissible.

* Female subjects who are pregnant or breast feeding.
* Clinical evidence (including physical exam, hemoglobin level and review of the medical history) of significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study.
* History of allergic reactions to ginseng, ginger, and Sichuan pepper.
* History of lactose intolerance.
* Subjects who are considered by the investigator to be alcoholics not in remission or known substance abusers.
* Subjects who have participated in another clinical study within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Gastric emptying of solid | 1 hr, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 8 hrs, 24 hrs, 48 hrs
Colonic geometric center at 24 hours | 4 hrs, 8 hrs, and 24 hrs
Ascending colon emptying | 1 hr, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 8 hrs, 24 hrs

SECONDARY OUTCOMES:
Colonic geometric center at 4 hours and 48 hours | 1 hr, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 8 hrs, 24 hrs, 48 hrs
Colonic filling at 6 hours | 1 hr, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs
Stool frequency | Day 1, Day 2, Day 3, Day 4, Day 5
Stool consistency | Day 1, Day 2, Day 3, Day 4, Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic, Rochester Methodist CRU
Locations (1):
- Mayo Clinic, Rochester Methodist CRU, Rochester, Minnesota, United States